CLINICAL TRIAL: NCT06218849
Title: Hybrid Interactive Avatars for Post-COVID Sufferers
Acronym: HINT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Cologne (Other)
Collaborators: University of Applied Sciences Cologne (Unknown); Humanizing Technologies GmbH (Unknown)
Responsible Party: Principal Investigator, Clara Lehmann, Prof. Dr. Clara Lehmann, University Hospital of Cologne
Other Study IDs: 16SV9183
Record Dates: First submitted 2024-01-22; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Post-COVID-19 syndrome; Avatar; App development
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate an app to improve communication and information flows for persons suffering from Post-COVID-19 syndrome (PCS). The main questions it aims to answer are:

* How can custom virtual characters (avatars) help to collect more data for the diagnosis of PCS?
* Can conversations with virtual (mobile) characters (avatars) and the presentation of health data help to improve the diagnosis and understanding of PCS?
* How should these virtual characters (avatars) be designed for people with PCS and healthcare professionals to be useful in the long term? This concerns appearance, dialog, personality and functions.

Participants will be asked to use and test the app and take part in two interviews at the beginning and end of the study.

DETAILED DESCRIPTION:
The overarching goal of the HINT project is to develop an app that people affected by PCS can use on their own devices in a language of their choice (e.g. their native language) to increase their health and data literacy about PCS and to provide socially equitable access to PCS care. Multilingual avatars are used for independent data collection, as the embodiment of interaction systems offers advantages for health queries. The data collected during the survey and - if desired - data from wearables are combined with historical data from the participants, processed and visualized. This allows patients to communicate with their avatar as well as with medical staff about their illness and its progression without language barriers affecting treatment. The avatar can also inform patients about new research findings on PCS. To this end, the system's level of knowledge is constantly compared with the current state of science; new findings are prepared for the target group and added to the knowledge base. The project is aimed at all those affected by PCS, although the multilingualism and low-threshold health education are intended to appeal in particular to people who have previously had difficulty accessing adequate care. The project is aimed at all those affected by PCS, although the multilingualism and low-threshold health education are intended to appeal in particular to people who have previously had difficulty accessing adequate care. The participatory and iterative development of the system, which also involves medical staff, contributes to overarching issues relating to co-creation approaches in the healthcare sector.

ELIGIBILITY:
Inclusion Criteria:

* Existence of a declaration of consent
* Stable clinical condition
* Diagnosis of Post-COVID syndrome according to the World Health Organization (WHO):

  * Symptoms persist for more than 12 weeks
  * Duration: at least 2 months
  * Etiology: no alternative diagnosis
  * Progression: persistent, recurrent, fluctuating

Exclusion Criteria:

* Known psychiatric or somatic illness that can explain the symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include female and male subjects who have been proven to have COVID-19 and are at least 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Final evaluation of the application field tests | 24 months after initiation of the study
  Following the successful completion of the field test (phase 2), a full evaluation will be carried out. The overall system and its use will be evaluated, taking into account both the perspective of those affected by PCS and that of the medical staff.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Cologne, Cologne, Northrhine-Westfalia, Germany